CLINICAL TRIAL: NCT01539239
Title: The Safety and Effectiveness of the Hydrus Aqueous Implant for Lowering Intraocular Pressure in Glaucoma Patients Undergoing Cataract Surgery, A Prospective, Multicenter, Randomized, Controlled Clinical Trial
Brief Title: Safety & Effectiveness Study of the Hydrus Microstent for Lowering IOP in Glaucoma Patients Undergoing Cataract Surgery (HORIZON)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivantis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP-11-001
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-02

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Glaucoma; POAG; Cataract
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrus Aqueous Implant (Treatment) (Experimental): Cataract surgery plus Hydrus Aqueous Implant
  Interventions: Device: Hydrus Aqueous Implant
- Cataract Surgery (Control) (Active Comparator): Cataract surgery only
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Device: Hydrus Aqueous Implant — The Hydrus Aqueous Implant is a crescent-shaped nitinol device intended to be a permanent implant placed through the trabecular meshwork into Schlemm's Canal, immediately following placement of a monofocal IOL.
  Arms: Hydrus Aqueous Implant (Treatment)
Procedure: Cataract surgery — A monofocal intraocular lens (IOL) placed during the cataract surgery.
  Arms: Cataract Surgery (Control)

SUMMARY:
This clinical trial is a prospective, randomized, controlled, multicenter, study. After informed consent is obtained, patients will be evaluated for eligibility based on glaucoma severity, eye health, and visual acuity. Following successful screening, use of all topical glaucoma medications will be stopped for a period of "washout" to establish a qualifying medication-free intraocular pressure (IOP) value. Clinical follow up will be scheduled over the course of the 24 month study, and examinations will be repeated to monitor eye health. At the 1 and 2 year follow up, those patients on ocular hypotensive medications will be instructed to washout, and then have the diurnal (IOP taken in the morning, mid-day, and afternoon in the same day) IOP evaluation. Annual follow up will occur up to 5 years. The primary effectiveness endpoint is a decrease in diurnal IOP from baseline compared to the 24 months diurnal IOP following medication washout.

ELIGIBILITY:
Inclusion Criteria:

* An operable age-related cataract
* A diagnosis of POAG treated with 1 to 4 hypotensive medications
* Medicated IOP ≤ 31 mmHg
* Diurnal IOP ≥ 22 mmHg and ≤ 34 mmHg

Exclusion Criteria:

* Congenital or developmental glaucoma
* Previous argon laser trabeculoplasty
* Ab-interno or ab-externo device implanted in or through Schlemm's Canal
* Use of oral hypotensive medication for glaucoma for treatment of fellow eye

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1143 (Actual)
Dates: Start 2012-01; Primary Completion 2017-06 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Crandall, MD, Principal Investigator — The Eye institute of Utah
Locations (38):
- United States (26):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Fayetteville, Arkansas
  - La Jolla, California
  - Orange, California
  - Sacramento, California
  - Fort Collins, Colorado
  - Parker, Colorado
  - Bradenton, Florida
  - Fort Myers, Florida
  - Ocala, Florida
  - Sioux City, Iowa
  - Garden City, Kansas
  - Louisville, Kentucky
  - Sandwich, Massachusetts
  - Bloomington, Minnesota
  - Chesterfield, Missouri
  - Wilmington, North Carolina
  - Cleveland, Ohio
  - Mason, Ohio
  - Maryville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Salt Lake City, Utah
  - Racine, Wisconsin
- Canada (2):
  - Edmonton, Alberta
  - Boisbriand, Quebec
- Mainz, Germany
- Parma, Italy
- Tijuana, Mexico
- Manila, Philippines
- Warsaw, Poland
- Spain (2):
  - Madrid
  - Zaragoza
- United Kingdom (3):
  - London
  - Manchester
  - Norwich

REFERENCES:
- [Derived] Zebardast N, Zheng C, Jampel HD. Effect of a Schlemm's Canal Microstent on Early Postoperative Intraocular Pressure after Cataract Surgery: An Analysis of the HORIZON Randomized Controlled Trial. Ophthalmology. 2020 Oct;127(10):1303-1310. doi: 10.1016/j.ophtha.2020.01.025. Epub 2020 Jan 23. PMID 32143828
- [Derived] Samuelson TW, Chang DF, Marquis R, Flowers B, Lim KS, Ahmed IIK, Jampel HD, Aung T, Crandall AS, Singh K; HORIZON Investigators. A Schlemm Canal Microstent for Intraocular Pressure Reduction in Primary Open-Angle Glaucoma and Cataract: The HORIZON Study. Ophthalmology. 2019 Jan;126(1):29-37. doi: 10.1016/j.ophtha.2018.05.012. Epub 2018 Jun 23. PMID 29945799

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened and enrolled at 38 investigational sites in the United States and other countries.
Pre-assignment Details: Of the 1,143 enrolled, 572 were screen failures and 15 were excluded intraoperatively due to failure to meet all intraoperative eligibility criteria. At the time of reporting, 556 patients randomized are available for analysis.
Period: Overall Study
Arm/Group | Hydrus Aqueous Implant (Treatment) | Cataract Surgery (Control)
Started | 369 | 187
Completed | 357 | 170
Not Completed | 12 | 17
Not completed — Death | 5 | 5
Not completed — Lost to Follow-up | 7 | 12

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) - All participants randomized and grouped according to their randomization assignment (as randomized). The ITT is used for the analyses of the primary and secondary effectiveness endpoints.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrus Aqueous Implant (Treatment) | Cataract Surgery (Control) | Total
Number analyzed (Participants) | 369 | 187 | 556
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (7.9) | 71.2 (7.6) | 71.1 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206 | 105 | 311
  Male | 163 | 82 | 245
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 19 | 43
  Not Hispanic or Latino | 345 | 168 | 513
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 11 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 45 | 15 | 60
  White | 291 | 153 | 444
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Mean Diurnal IOP From Baseline at 24 Months Following Medication Washout.
Description: Percentage of eyes in which diurnal IOP was reduced by greater than or equal to 20% at 24 months postoperative compared to baseline after washout of topical glaucoma medications.
Time Frame: Baseline and 24 months
Population: Intent-to-Treat (ITT)
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Hydrus Aqueous Implant (Treatment) | Cataract Surgery (Control)
Number analyzed (Participants) | 369 | 187
Number analyzed (Eyes) | 369 | 187
percentage of eyes | 77.2 | 57.8

2. Secondary Outcome: Mean Diurnal Washed Out IOP Change From Baseline at 24 Months Compared Between Treatment and Control Groups.
Description: Mean diurnal IOP change from baseline at 24 months between both groups after washout of topical glaucoma medications.
Time Frame: Baseline and 24 months
Population: Intent-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hydrus Aqueous Implant (Treatment) | Cataract Surgery (Control)
Number analyzed (Participants) | 369 | 187
mmHg | -7.5 (4.1) | -5.3 (3.9)

ADVERSE EVENTS:
Time Frame: 24 months
Description: An adverse event is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the investigational medical device. All subjects who have been exposed to the study treatment were evaluated for adverse events.
Arm/Group | Hydrus Aqueous Implant (Treatment) | Cataract Surgery (Control)
All-Cause Mortality (participants affected / at risk) | 5/369 | 5/187
Serious Adverse Events (participants affected / at risk) | 10/369 | 6/187
Other Adverse Events (participants affected / at risk) | 106/369 | 24/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrus Aqueous Implant (Treatment) (N=369) | Cataract Surgery (Control) (N=187)
BCVA loss greater than or equal to 2 lines ETDRS greater than or equal to 3 months (Eye disorders) | 0 (0) | 1 (1)
Corneal Edema Mild to Mod after 1 month (Eye disorders) | 1 (1) | 0 (0)
Glaucoma progression (Eye disorders) | 0 (0) | 1 (1)
Neovascular Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Repair of malpositioned IOL haptic (Eye disorders) | 1 (1) | 0 (0)
Orbital hemangioma (Eye disorders) | 1 (1) | 0 (0)
Squamous cell carcinoma of the conjunctiva (Eye disorders) | 1 (1) | 0 (0)
Worsening of visual field MD by greater than or equal to 2.5 dB compared with preoperative (Eye disorders) | 0 (0) | 1 (1)
Retinal Complications (Eye disorders) | 6 (6) | 4 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrus Aqueous Implant (Treatment) (N=369) | Cataract Surgery (Control) (N=187)
Anterior uveitis/iritis (non-persistent) (Eye disorders) | 19 (19) | 3 (3)
Conjunctivitis (Eye disorders) | 21 (27) | 13 (14)
Device obstruction, partial or complete (Eye disorders) | 27 (27) | 0 (0)
Peripheral anterior synechiae without device obstruction (Eye disorders) | 27 (27) | 0 (0)
Worsening of visual field MD by greater than or equal to 2.5 dB compared with preoperative (Eye disorders) | 16 (16) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sites participating in the trial may not publish their single center results until the aggregate study results have been published unless first obtaining written consent from the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-11-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT01539239/Prot_SAP_000.pdf